CLINICAL TRIAL: NCT00448383
Title: An Open-Label, Multi-Center Study to Assess the Safety and Efficacy of the Fully Human Anti-TNF-α Monoclonal Antibody Adalimumab (D2E7) When Added to Inadequate Standard Anti-Rheumatic Therapy in Patients With Active Rheumatoid Arthritis
Brief Title: A Study to Assess the Safety and Efficacy of Adalimumab When Added to Inadequate Standard Anti-Rheumatic Therapy in Patients With Active Rheumatoid Arthritis
Acronym: ReAct
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Larry McNamee, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-497
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

ARMS (1):
- 1 (Experimental): Open-label adalimumab
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — 40mg every other week
  Other Names: ABT-D2E7; Humira

SUMMARY:
This is an open-label, multi-center study in which adalimumab (D2E7) is administered subcutaneously 40 mg every other week in addition to current anti-rheumatic therapies. Patients must have active disease despite standard anti-rheumatic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years or older
* ACR criteria for diagnosis of RA for at least 3 months.
* Active RA as defined by DAS28 >= 3.2 at study entry.
* Unsatisfactory response or intolerance to prior DMARDs.
* A negative pregnancy test (serum HCG) for women of childbearing potential prior to start of study treatment.
* Use of reliable method of contraception e.g. IUDs, condoms, or hormone (oral, implantable, or injectable) contraceptives by all female patients of childbearing potential. Male patients with procreative capacity should also ensure that effective contraception is used during the study and for 70 days after study completion

Exclusion Criteria:

* Prior treatment with alkylating agents such as cyclophosphamide or chlorambucil.
* Prior treatment with intravenous immunoglobulin or any investigational agent within 30 days, or 5 half lives of the product, whichever is longer.
* Prior treatment with investigational biologic therapy (e.g. anti CD4)
* Treatment within the last 2 months with approved biologic therapy (eg etanercept, infliximab, anakinra)
* Prior treatment with total lymphoid irradiation
* History of cancer or lymphoproliferative disease other than a successfully and completely treated squamous cell or basal cell carcinoma.
* History of or current acute inflammatory joint disease of origin other than RA, e.g. mixed connective tissue disease, systemic lupus erythematosus etc.
* History of uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent stroke (within 3 months) and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
* Positive serology for hepatitis B or C indicating active infection
* History of positive HIV status.
* Persistent infection, or severe infections requiring hospitalization or treatment with iv antibiotics within 30 days, or oral antibiotics within 14 days prior to enrollment.
* Female subjects who are pregnant or breast-feeding.
* History of clinically significant drug or alcohol abuse in the last year.
* Previous diagnosis or signs of demyelinating diseases
* History of active tuberculosis (TB), histoplasmosis or listeriosis.
* Signs of previous TB infection (chest X-ray signs or positive PPD skin test). The diagnosis of previous TB infection will be based on chest X-ray signs and on PPD skin test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6610 (Actual)
Dates: Start 2002-09; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Change of disease activity score (DAS28) compared with study entry | Week 12
EULAR and ACR response criteria at week 12 | Week 12

SECONDARY OUTCOMES:
Adverse events | Baseline - Week 12
Clinical laboratory parameters | Screening, Week 6 & Week 12 and/or ET

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778
- [Derived] Burmester GR, Matucci-Cerinic M, Mariette X, Navarro-Blasco F, Kary S, Unnebrink K, Kupper H. Safety and effectiveness of adalimumab in patients with rheumatoid arthritis over 5 years of therapy in a phase 3b and subsequent postmarketing observational study. Arthritis Res Ther. 2014 Jan 27;16(1):R24. doi: 10.1186/ar4452. PMID 24460746
- [Derived] Burmester GR, Ferraccioli G, Flipo RM, Monteagudo-Saez I, Unnebrink K, Kary S, Kupper H. Clinical remission and/or minimal disease activity in patients receiving adalimumab treatment in a multinational, open-label, twelve-week study. Arthritis Rheum. 2008 Jan 15;59(1):32-41. doi: 10.1002/art.23247. PMID 18163417